CLINICAL TRIAL: NCT02224040
Title: Typhoid Fever: Combined vs. Single Antibiotic Therapy. A Prospective Randomized Controlled Study in Nepal.
Brief Title: Typhoid Fever: Combined vs. Single Antibiotic Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Eli Schwartz MD, DTMH, Principal Investigator of the geographic clinical, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64/12
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever | interventions — Ceftriaxone; Azithromycin; Cefixime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ceftriaxone I.V (Experimental): The participants in this arm will receive the following drug and dosage: adult: Ceftriaxone intravenous 2 gr once a day. Pediatric: intravenous 75 mg/kg ceftriaxone once a day (maximum dose 2.5 g/day). Patients will receive antibiotic treatment until defervescence and for 3 days afterwards. Patients will be hospitalized during the entire treatment course (including the afebrile period).
  Interventions: Drug: ceftriaxone
- Ceftriaxone I.V+Azithromycin P.O (Experimental): The participants in this arm will receive the following drugs and dosages: adult: 2 g intravenous ceftriaxone and 500 mg oral azithromycin once a day. Pediatric: intravenous 75 mg/kg ceftriaxone once a day and oral 20 mg/kg azithromycin suspension once a day. Patients will receive antibiotic treatment until defervescence and for 3 days afterwards. Patients will be hospitalized during the entire treatment course (including the afebrile period).
  Interventions: Drug: ceftriaxone and azithromycin
- Azithromycin P.O (Experimental): The participants in this arm will receive the following drug and dosage: adult: azithromycin oral 500 mg once a day. Pediatric: oral 20 mg/kg azithromycin suspension once a day (maximum dose 1000 mg/day). Patients will receive antibiotic treatment until defervescence and for 3 days afterwards.
  Interventions: Drug: azithromycin
- Azithromycin P.O+Cefixime P.O (Experimental): The participants in this arm will receive the following drugs and dosages: adult: 500 mg azithromycin and 400 mg cefixime. Pediatric: oral 20 mg/kg azithromycin suspension once a day and oral 10 mg/kg cefixime. Patients will receive antibiotic treatment until defervescence and for 3 days afterwards.
  Interventions: Drug: azithromycin and cefixime

INTERVENTIONS:
Drug: ceftriaxone
  Arms: Ceftriaxone I.V
Drug: ceftriaxone and azithromycin
  Arms: Ceftriaxone I.V+Azithromycin P.O
Drug: azithromycin
  Arms: Azithromycin P.O
Drug: azithromycin and cefixime
  Arms: Azithromycin P.O+Cefixime P.O

SUMMARY:
The current study goal is to examine the effect of Cephalosporins, Azithromycin and the combination of both on typhoid fever therapy in endemic population.

The investigator's hypothesize that the combination of azithromycin and ceftriaxone may prove superior to each drug, ceftriaxone or azithromycin, alone.

DETAILED DESCRIPTION:
Typhoid Fever is a highly prevalent infection in the Indian subcontinent. Due to multidrug resistant strains in these areas, third generation cephalosporins, such as ceftriaxone, are the treatment of choice. However, the latter regimen exhibits a slow response with mean time of 5 to 7 days or even longer to defervescence, which could be attributed to poor penetration capability of the drug into cells, and thus difficulty to eradicate the bacteria from the intracellular niche.

Attempts have been made to overcome this setback by introducing alternative antibiotic regimens, such as azithromycin. However studies comparing between azithromycin and a third-generation cephalosporin for the treatment of typhoid fever in adult population in the Indian subcontinent are lacking.

Over the last few years our approach towards non-immunized travelers, who acquired typhoid fever in the Indian subcontinent, was to administer a combination therapy of intravenous ceftriaxone with oral azithromycin. The rationale of this dual regimen was its pharmacokinetic profile, which suggests a complimentary action of the two agents - ceftriaxone on the extracellular compartment and azithromycin on the intracellular compartment. Moreover, in our clinical experience, preliminary published data has proven combination therapy significantly superior to ceftriaxone alone albeit in a small group of travelers.

In the current study the investigators intend to compare the efficacy of ceftriaxone vs. azithromycin and vs. combined therapy of both agents for the treatment of uncomplicated typhoid fever in terms of time to defervescence.

4 different treatment strategies will be examined (as mentioned in the arm section). All participants will be checked for vital signs, will undergo physical examination, ECG, laboratory testing, blood, urine and stool culture and tests for susceptibility to antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Blood culture-proven typhoid fever (S. typhi or S. paratyphi)
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Allergy to ceftriaxone or macrolides
* Major typhoid fever-associated complications
* Inability to swallow oral medication
* Underlying illness
* Pregnancy
* Lactation
* Treatment within the past 4 days with an antibiotic that may be effective against typhoid fever

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Fever clearance time | One month
  Time to fever clearance will be measured and will be defined as an oral temperature that is below 37.50 C

SECONDARY OUTCOMES:
Treatment failure | One month
  Secondary endpoints will be treatment failure (defined as the need to switch antibiotic treatment according to physician's decision such as high grade fever after 5 days of treatment, appearance of typhoid complications under the treatment), clearance of bacteremia, development of typhoid-related complications, late relapse, fecal carriage and adverse drug reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Schwartz, MD, DTMH, Principal Investigator — Sheba Medical Center
Locations (1):
- Dhulikhel hospital, Dhulikhel, Nepal

REFERENCES:
- [Derived] Zmora N, Shrestha S, Neuberger A, Paran Y, Tamrakar R, Shrestha A, Madhup SK, Bedi TRS, Koju R, Schwartz E. Open label comparative trial of mono versus dual antibiotic therapy for Typhoid Fever in adults. PLoS Negl Trop Dis. 2018 Apr 23;12(4):e0006380. doi: 10.1371/journal.pntd.0006380. eCollection 2018 Apr. PMID 29684022